CLINICAL TRIAL: NCT04275765
Title: Community Enabled Readiness for First 1000 Days Learning Ecosystem
Acronym: CRADLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Ng Kee Chong, Senior Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201907-00050
Record Dates: First submitted 2020-01-20; First posted 2020-02-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Emotional Well-being of First-time Families; Nutritional Health of Mother and Child; Parenting Self-Efficacy for First-time Families; Experience of First-time Families

STUDY DESIGN:
Intervention Model Description: Interventional study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Routine Care (No Intervention): Participants will undergo routine care but take part in assessments.
- Arm 2:Behavioral Intervention with nudges & Facebook (Active Comparator): Participants will receive nudges and be enrolled in social media platform.
  Interventions: Behavioral: Arm 2:Behavioral Intervention with nudges & Facebook interaction
- Arm 3: Community Intervention with individualised teleconferencing sessions and phone calls. (Active Comparator): Participants will receive individualised teleconferencing sessions and phone calls by skilled midwives.
  Interventions: Other: Arm 3: Community Intervention with individualised teleconferencing sessions and phone calls.

INTERVENTIONS:
Behavioral: Arm 2:Behavioral Intervention with nudges & Facebook interaction — Participants will receive nudges and be enrolled to Facebook group for self-learning.
  Arms: Arm 2:Behavioral Intervention with nudges & Facebook
Other: Arm 3: Community Intervention with individualised teleconferencing sessions and phone calls. — Participants will receive individualised teleconferencing sessions and phone calls by skilled midwives.
  Arms: Arm 3: Community Intervention with individualised teleconferencing sessions and phone calls.

SUMMARY:
The CRADLE (Community-enabled Readiness-for-1000-Days Learning Ecosystem) initiative seeks to improve first-time families' self-efficacy in parenting and to tangibly impact factors in maternal and child care which will result in improved health of mother and child.

DETAILED DESCRIPTION:
Title: CRADLE (Community enabled Readiness for first 1000-Days Learning Ecosystem) Project

Introduction:

The "developmental origins of health and disease" (DOHaD) is a concept that has emerged over the past 50 years, linking the state of health and risk from disease in early childhood and adult life. With increasing evidence in neuroscience of the critical window of the first 1000 days of life which has life- long impact on cognitive, behavioral, physical and mental health of an individual. In present society where new parents learned the skills from social media which are based on personal perception and not evidence.

CRADLE (Community-enabled Readiness-for-1000-Days Learning Ecosystem) initiative seeks to improve first-time families' self-efficacy in parenting and to tangibly impact factors in maternal and child care which will result in improved health of mother and child.

Hypothesis:

Use of an integrated choice architecture in a self-learning eco-community, with calibrated nudges, and group interactions & interaction with midwives and individualised teleconferencing sessions in the first 1000-days for first-time families will improve parenting self-efficacy.

Method:

This will be an Interventional Cohort Study. Each ARM 250 subjects. ARM 1 : Routine care ARM 2 : Behavioral Intervention with nudges and Facebook interaction ARM 3 : Community Intervention with interaction with midwives and individualised teleconferencing sessions

The follow up period will be from first contact till child reaches 2 years old Measurement.

The investigators will quantify the impact of this initiative through measurements of specific health & nutrition domains & patient-reported outcome measures (see below) as well as participant satisfaction.

The two key health morbidities the investigators are addressing are the overall health and mental wellness of first-time families as well as their metabolic health (ie, nutrition).

1. Mother's Height and Weight (BMI)
2. Child's Height and Weight (BMI)
3. PROMIS Global-10 Scale
4. Patient Health Questionaire-2
5. Edinburgh Postnatal Depression Scale
6. Parental Sense Of Competency Scale
7. Tool To Measure Parenting Self-Efficacy (TOPSE)
8. Birth Satisfaction Scale
9. Breastfeeding Self-Efficacy Scale
10. Infant Feeding Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. First-time mothers
2. Be at least 17 years of age
3. Is residing in Singapore for the next 3 years
4. Understand English, or has a family member who is able to assist.

Exclusion Criteria:

1. Has existing medical conditions such as chronic illnesses

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — First-time mothers
Enrollment: 750 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Parenting self-efficacy | Up to 24 months of age, from 6 weeks after birth until 24 months of age
  Parenting self-efficacy as assessed by the Tool to measure Parenting Self-Efficacy, which is domain-specific.
Parenting self-efficacy | Up to 24 months of age, from 6 weeks after birth until 24 months of age
  Parenting self-efficacy as assessed by the Parental Sense of Competence Scale, which is domain-general.

SECONDARY OUTCOMES:
Health experience | Up to 18 months of age, from first trimester in pregnancy until 18 months during the postnatal period
  Health Experience as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global10.
Birth experience | At point of birth
  Birth Experience as assessed by the Birth Satisfaction Scale - Revised.
Mental wellness | Up to 6 months of age, from first trimester in pregnancy up to 6 months during postnatal period
  Mental wellness as assessed by the Patient Health Questionnaire-2.
Depressive symptoms | Up to 6 months of age, from first trimester in pregnancy up to 6 months during postnatal period
  Depressive symptoms as assessed by the Edinburg Postnatal Depression Scale (EPDS).
Maternal nutritional status | Through study completion, from first trimester in pregnancy up to 24 months during postnatal period
  Maternal nutritional status as assessed based on weight status, i.e. weight gain and weight retention.
Child nutritional status | From birth until up to 24 months during postnatal period
  Child nutritional status as assessed based on weight and height.
Breastfeeding self-efficacy | From birth until up to 6 months during postnatal period
  Breastfeeding self-efficacy as assessed by the Breastfeeding Self-Efficacy Score-Short Form.
Maternal feeding beliefs and practices | At 18 months of age, at 18 months during postnatal period
  Maternal feeding beliefs and practices as assessed by the Infant Feeding Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kee Chong Ng, MMed, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Access to IPD will be limited to the project study team only.

REFERENCES:
- [Derived] Loy SL, Thilagamangai, Teo J, Chan SW, Razak NKA, Chay OM, Ng KC. A Community-enabled Readiness for first 1000 Days Learning Ecosystem (CRADLE) for first-time families: study protocol of a three-arm randomised controlled trial. Trials. 2021 Mar 6;22(1):191. doi: 10.1186/s13063-021-05144-5. PMID 33676560
- See also: PROMIS GLOBAL HEALTH — https://www.codetechnology.com/promis-global-10/
- See also: THE PATIENT HEALTH QUESTIONAIRE-2 (PHQ-2) — http://www.systematicreviewsjournal.com/content/3/1/124
- See also: EDINBURGH POSTNATAL DEPRESSION SCALE (EPDS) — https://www.ncbi.nlm.nih.gov/pubmed/3651732
- See also: PARENTAL SENSE OF COMPETENCY SCALE (PSOC) — https://www.bristol.ac.uk/media-library/sites/sps/documents/c-change/parenting-sense-of-competence-scale.pdf
- See also: TOPSE Tool to measure Parenting Self-Efficacy — https://www.topse.org.uk/site/what-is-topse/
- See also: BREASTFEEDING SELF-EFFICACY SCORE- SHORT FORM — https://www.ncbi.nlm.nih.gov/pubmed/14649593
- See also: BIRTH SATISFACTION SCALE-REVISED — https://www.ncbi.nlm.nih.gov/pubmed/21456488
- See also: INFANT FEEDING QUESTIONNAIRE — https://www.ncbi.nlm.nih.gov/pubmed/11773804